CLINICAL TRIAL: NCT01129011
Title: 6-Month, Phase 3, Randomized, Double-blind, Parallel-group, Controlled, Multi-center Study Evaluate Gastric Ulcer Incidence Following Administration of PN400 or Naproxen in Subjects Who Are at Risk for Developing NSAID-associated Ulcers
Brief Title: Evaluating PN 400 (VIMOVO) in Reducing Gastric Ulcers Compared to Non-steroidal Antiinflammatory Drug (NSAID) Naproxen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Senior Vice President, Clinical Research, Pozen, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN400-302
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-11

CONDITIONS: Gastric Ulcer
Keywords: NSAID; gastric ulcers; Vimovo; Esomeprazole; Naproxen
MeSH Terms: conditions — Stomach Ulcer | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PN400 (Experimental): Naproxen 500 mg/Immediate-Release Esomeprazole 20 mg dosed twice daily
  Interventions: Drug: PN400 (VIMOVO)
- Naproxen (Active Comparator): Naproxen 500 mg dosed twice daily
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: PN400 (VIMOVO) — PN400 tablets (Naproxen 500 mg and Esomeprazole 20 mg) twice daily (bid) taken orally.
  Other Names: Vimovo
  Arms: PN400
Drug: Naproxen — Naproxen 500 mg dosed twice daily (bid) orally
  Other Names: Naprosyn
  Arms: Naproxen

SUMMARY:
This study uses a randomized, double-blind, controlled design to demonstrate that PN400 (esomeprazole and naproxen) is more effective in reducing the occurrence of gastroduodenal ulcers, dyspepsia, and heartburn in subjects at risk for developing NSAID-associated gastric ulcers compared to naproxen alone.

DETAILED DESCRIPTION:
Objectives:

Primary: To demonstrate that PN400 is effective in reducing the risk of gastric ulcers in subjects at risk for developing NSAID-associated gastric ulcers.

Secondary:

* To determine if PN400 is effective in reducing the risk of duodenal ulcers in subjects at risk for developing NSAID-associated ulcers
* To compare upper gastrointestinal symptoms in subjects treated with PN400 versus naproxen as measured by scores on the Severity of Dyspepsia Assessment (SODA) instrument and the Overall Treatment Evaluation - Dyspepsia (OTE-DP)
* To compare heartburn symptoms in subjects treated with PN400 versus naproxen
* To evaluate the safety and tolerability of PN400 and naproxen

ELIGIBILITY:
Inclusion Criteria

A subject was eligible for inclusion in this study if all of the following criteria applied:

1. Male or non-pregnant, non-breastfeeding female subjects with a history of osteoarthritis, rheumatoid arthritis, ankylosing spondylitis or other medical conditions expected to require daily NSAID therapy for at least 6 months, who were

   * 18-49 years of age and had a history of a documented, uncomplicated gastric or duodenal ulcer (a mucosal break of at least 3 mm in diameter with depth, without any concurrent bleeding, clot or perforation) within the past 5 years OR, who were
   * 50 years of age and older (These subjects did not require a history of a documented, uncomplicated gastric or duodenal ulcer within the past 5 years.)
2. Female subjects were eligible for participation in the study if they were of

   * non-childbearing potential (i.e., physiologically incapable of becoming pregnant);
   * childbearing potential, had a negative pregnancy test at Screening, and at least 1 of the following applied or was agreed to by the subject:
   * Female sterilization or sterilization of male partner
   * Hormonal contraception by oral route, implant, injectable, vaginal ring
   * Any intrauterine device with published data showing that the lowest expected failure rate is < 1% per year
   * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide)
   * Any other method with published data showing that the lowest expected failure rate is < 1% per year
3. Each subject was required to understand and comply with study procedures required of a subject and was able and willing to provide written informed consent prior to any study procedures being performed.

Exclusion Criteria

A subject was not eligible for this study if any 1 or more of the following criteria applied:

1. History of hypersensitivity to esomeprazole or to another PPI
2. History of allergic reaction or intolerance to any NSAID (including aspirin) and/or a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps
3. Participation in any study of an investigational treatment in the 4 weeks before Screening
4. Presence of uncontrolled acute or chronic medical illness, e.g., GI disorder, hypertension, diabetes, thyroid disorder, depression and/or infection that would have endangered a subject if they were to have participated in the study
5. GI disorder or surgery leading to impaired drug absorption
6. Evidence of uncontrolled, or unstable cardio- or cerebrovascular disorder, which in the investigator's opinion would have endangered a subject if they were to have participated in the study
7. Schizophrenia or bipolar disorder
8. Use of any excluded concomitant medication (see Section 9.4.8)
9. A recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence, including overuse/abuse of narcotics for management of pain
10. Serious blood coagulation disorder, including use of systemic anticoagulants
11. Positive test result for H. pylori at Screening
12. Screening endoscopy showing any gastric or duodenal ulcer at least 3 mm in diameter with depth
13. Screening laboratory alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value > 2 times the upper limit of normal
14. Estimated creatinine clearance < 30 ml/min
15. Other than noted specifically, any screening laboratory value that was clinically significant in the investigator's opinion and would have endangered a subject if they were to have participated in the study
16. History of malignancy, treated or untreated, within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everardus Orlemans, PhD, Study Chair — POZEN

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center US study in which 70 sites recruited subjects between September 2007 and September 2008
Pre-assignment Details: Screening for eligibility and wash-out of restricted medications
Groups:
- PN400 (VIMOVO): Naproxen 500 mg/Immediate-Release Esomeprazole 20 mg dosed twice daily (bid)
- Naproxen: Naproxen 500 mg dosed twice daily (bid)
Period: Overall Study
Arm/Group | PN400 (VIMOVO) | Naproxen
Started | 210 (Safety, Intent-to-Treat population) | 210 (Safety, Intent-to-Treat population)
Completed | 151 | 153
Not Completed | 59 | 57
Not completed — Adverse Event | 20 | 30
Not completed — Withdrawal by Subject | 24 | 8
Not completed — Lost to Follow-up | 6 | 7
Not completed — Duodenal Ulcer | 2 | 8
Not completed — misc | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PN400 (VIMOVO) | Naproxen | Total
Number analyzed (Participants) | 210 | 210 | 420
Age Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.2) | 59.4 (8.3) | 59.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 142 | 274
  Male | 78 | 68 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gastric Ulcer Confirmed by Endoscopy
Description: The primary efficacy endpoint was the number of subjects with gastric ulcers at any time throughout 6 months of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter (measured by close application of open endoscopic biopsy forceps) with unequivocal crater depth. A subject is considered to have completed the study if all scheduled assessments up through the 6 month visit have been performed or if the endpoint of gastric ulcer confirmed by endoscopy has been reached.
Time Frame: 6 months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: Participants
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Participants | 15 [4.1 to 11.5] | 51 [18.6 to 30.7]
Statistical Analysis 1: Comparison: PN400 (VIMOVO) vs Naproxen; The primary efficacy endpoint was the proportion of subjetcs developing gastric ulcers throughout 6 months of study treatment. A summary, including cumulative frequency and percentage with associated 95% confidence intervals was produced for the observational incidences of gastric ulcers at 6 months. The cumulative proportion of subjects developing gastric ulcers at 6 months was analyzed using the CMH test stratified by use of low-dose aspirin (Yes/No) at randomization; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; CMH test stratified by use of low-dose aspirin (Yes/No) at randomization; proportions = 11.9, 95% CI 2-sided [7.9 to 17.1]

2. Secondary Outcome: The Number of Participants With Pre-Specified NSAID-Associated Upper GI Adverse Events or Duodenal Ulcers
Description: The Number of Participants with Pre-Specified non-steroidal antiinflammatory drug (NSAID)-Associated Upper Gastrointestinal (UGI) Adverse Events or Duodenal Ulcers after 6 months of treatment. Pre-specified UGI adverse events typically associated with NSAID use include dyspepsia, abdominal pain, gastritis, erosive esophagitis, duodenitis, abdominal discomfort
Time Frame: 6 months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: Participants
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Participants | 114 [47.3 to 61.2] | 151 [65.3 to 77.9]
Statistical Analysis 1: Comparison: PN400 (VIMOVO) vs Naproxen; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: The Number of Participants Discontinuing From the Study Due to NSAID-Associated Upper GI Adverse Events or to Duodenal Ulcer
Description: The Number of Participants Discontinuing from the Study Due to non-steroidal antiinflammatory drug (NSAID)-Associated Upper GI Adverse Events or to Duodenal Ulcer during the treatment period
Time Frame: 6 Months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: Participants
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Participants | 10 [2.3 to 8.6] | 25 [7.9 to 17.1]
Statistical Analysis 1: Comparison: PN400 (VIMOVO) vs Naproxen; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel

4. Secondary Outcome: The Number of Participants Developing Duodenal Ulcers Throughout 6 Months of Treatment
Description: The Number of Participants Developing Duodenal Ulcers at any time during the 6 Months of the treatment period
Time Frame: 6 months
Population: Intent to treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Participants | 2 [0.1 to 3.4] | 12 [3.0 to 9.8]
Statistical Analysis 1: Comparison: PN400 (VIMOVO) vs Naproxen; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel

5. Secondary Outcome: Heartburn Symptom Resolution, ie no Heartburn Symptoms During the Last 7 Days Prior to the Visit
Description: Subjects were asked whether heartburn symptoms within the 7 days prior to the visit were:
  * none: no symptoms
  * mild: awareness of symptom, but easily tolerated
  * moderate: discomforting symptom sufficient to cause interference with normal activities (including sleep)
  * severe: incapacitating symptom, with inability to perform normal activities (including sleep) Heartburn was defined as a burning feeling rising from the stomach or lower part of the chest towards the neck.
Time Frame: 6 months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
participants | 102 | 62
Statistical Analysis 1: Comparison: PN400 (VIMOVO) vs Naproxen; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Improvement From Baseline in Upper Abdominal Pain and Discomfort Scores at 6 Months, Based on the Overall Treatment Evaluation for Dyspepsia Questionnaire
Description: Improvement from baseline in Upper Abdominal Pain and Discomfort scores at 6 months, based on the overall Treatment Evaluation for Dyspepsia Questionnaire. Subjects were asked: "since treatment started, has there been any change in your upper abdominal pain and/or discomfort?" Answers would be better/about the same/worse. Participants with the response "better" (instead of "about the same" or "worse"), are tabulated by treatment group.
Time Frame: change from baseline at 6 Months
Population: Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Participants | 79 | 63

7. Secondary Outcome: Mean Change From Baseline on Pain Intensity of the Severity of Dyspepsia Assessment (SODA) Subscales
Description: Mean Change from Baseline on Pain Intensity of the Severity of Dyspepsia Assessment (SODA) Subscales. There are 6 questions about abdominal pain during the past 7 days: q 1-5 on average: 1. rate with a number between 0 (no pain) and 100 (pain as bad as it could be), 2. rate with a number between 0 (no discomfort) and 10 (discomfort as bad as it can be), 3. on a scale of 5 (from none to excriciating), 4. on 100 mm VAS, 5. on a scale of 4 and 6. worst abdominal pain scale 0 (no discomfort) and 10 (discomfort as bad as it can be). Total composite possible range for "pain intensity" is: 2-47
Time Frame: Baseline to 6 Months
Population: Intent to Treat (ITT) Population
Measure: Least Squares Mean (Standard Error); unit: Units on SODA Subscale
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Units on SODA Subscale | -3 (0.7) | 0 (0.7)

8. Secondary Outcome: Mean Change From Baseline on Non-Pain Symptoms of the Severity of Dyspepsia Assessment (SODA) Subscales
Description: Change from Baseline of Non-Pain Symptoms on the SODA Assessment. There are 7 categories about the non-pain symptoms: burping/beching, heartburn, bloating, passing gas, sour taste, nausea and bad breath. For each of these categories, subjects were to rate during the past seven days, on average, the severity on a 5 point scale ranging from no problem to very severe problem. The scores are combined into a single composite score. The total possible range of the non-pain symptoms subscale is: 7-35.
Time Frame: baseline to 6 Months
Population: Intent to Treat (ITT) Population
Measure: Least Squares Mean (Standard Error); unit: Units on SODA Subscale
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Units on SODA Subscale | -1.1 (0.3) | 0.1 (0.3)

9. Secondary Outcome: Mean Change From Baseline on Satisfaction of the Severity of Dyspepsia Assessment (SODA) Subscales
Description: Mean Change in Satisfaction on SODA Assessment. Questions/statements to rate about satisfaction/dissatisfaction with their present level of abdominal discomfort. Question 1: 4-point scale range 0 (extremely unhappy) to 4 (extremely happy), statement 2 (I feel satisfied with my health with regard to abdominal discomfort) & statement 3 (I am pleased because my abdominal discomfort seems under control) on a 5 point scale (definitely true to definitely false) & question 4 rated how pleased subjects were with abdominal discomfort on a 10 point scale. Total satisfaction composite range: 2-23
Time Frame: baseline to 6 Months
Population: Intent to Treat (ITT) Population
Measure: Least Squares Mean (Standard Error); unit: Units on SODA Subscale
Arm/Group | PN400 (VIMOVO) | Naproxen
Number analyzed (Participants) | 210 | 210
Units on SODA Subscale | 1.9 (0.4) | 0.5 (0.4)

ADVERSE EVENTS:
Time Frame: Randomization through 6 months
Arm/Group | PN400 (VIMOVO) | Naproxen
Serious Adverse Events (participants affected / at risk) | 5/210 | 7/210
Other Adverse Events (participants affected / at risk) | 160/210 | 174/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN400 (VIMOVO) (N=210) | Naproxen (N=210)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Post-procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN400 (VIMOVO) (N=210) | Naproxen (N=210)
Dyspepsia (Gastrointestinal disorders) | 41 (41) | 49 (49)
Gastritis erosive (Gastrointestinal disorders) | 38 (38) | 81 (81)
Gastritis (Gastrointestinal disorders) | 34 (34) | 32 (32)
Abdominal pain upper (Gastrointestinal disorders) | 15 (15) | 19 (19)
Nausea (Gastrointestinal disorders) | 13 (13) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 9 (9)
Hiatus hernia (Gastrointestinal disorders) | 10 (10) | 11 (11)
Oesophagitis (Gastrointestinal disorders) | 8 (8) | 15 (15)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (5)
Flatulence (Gastrointestinal disorders) | 7 (7) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 6 (6)
Erosive duodenitis (Gastrointestinal disorders) | 5 (5) | 20 (20)
Abdominal pain lower (Gastrointestinal disorders) | 4 (4) | 7 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 8 (8)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 12 (12)
Erosive oesophagitis (Gastrointestinal disorders) | 2 (2) | 12 (12)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 8 (8)
Sinusitis (Infections and infestations) | 5 (5) | 6 (6)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Dysgeusia (Nervous system disorders) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that the first publication will be a multi-center publication of the study results. Following this multi-center publication, PI can publish, present or use any non-confidential study results following Sponsor review and comment.